CLINICAL TRIAL: NCT04570436
Title: A Phase 4, Randomized, Double-blind, Double-dummy, Placebo and Active-controlled, Single-dose, Five-way Crossover Study Evaluating the Abuse Potential of Three Doses of NEURONTIN® Taken Orally in Healthy, Non-drug Dependent Participants With Sedative Drug Abuse Experience
Brief Title: Evaluating the Abuse Potential of NEURONTIN® When Taken Orally in Healthy Non-drug Dependent Participants With Sedative Drug Abuse Experience
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Viatris Specialty LLC (Industry)
Responsible Party: Sponsor
Organization: Viatris Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: A9451181
Record Dates: First submitted 2020-09-24; First posted 2020-09-30 (Actual); Results first posted 2023-12-06 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Abuse Potential
Keywords: Neurontin; Diazepam; Abuse Liability; Gabapentin
MeSH Terms: interventions — Gabapentin; Diazepam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- gabapentin 600 mg (Experimental): single dose
  Interventions: Drug: gabapentin 600 mg
- diazepam 20 mg (Active Comparator): single dose
  Interventions: Drug: diazepam 20 mg
- placebo (Placebo Comparator): single dose
  Interventions: Other: placebo
- gabapentin 1200 mg (Experimental): single dose
  Interventions: Drug: gabapentin 1200 mg
- gabapentin 1800 mg (Experimental): single dose
  Interventions: Drug: gabapentin 1800 mg

INTERVENTIONS:
Drug: gabapentin 600 mg — participants will receive an oral dose of gabapentin 600 mg
  Arms: gabapentin 600 mg
Drug: gabapentin 1200 mg — participants will receive an oral dose of gabapentin 1200 mg
  Arms: gabapentin 1200 mg
Drug: gabapentin 1800 mg — participants will receive an oral dose of gabapentin 1800 mg
  Arms: gabapentin 1800 mg
Drug: diazepam 20 mg — participants will receive an oral dose of 20 mg dose of diazepam
  Arms: diazepam 20 mg
Other: placebo — participants will receive an oral dose of placebo
  Arms: placebo

SUMMARY:
This will be a randomized, double-blind, double-dummy, placebo- and active controlled, 5 treatment, 10 sequence, 5 period crossover single dose, Williams square design study in healthy adult, non drug dependent male and female participants with drug abuse experience with sedative drugs.

DETAILED DESCRIPTION:
The study includes Screening, a Qualification Phase consisting of a Naloxone Challenge and Drug Discrimination crossover study, a Treatment Phase and Follow-up. Following successful completion of the Qualification Phase the participants will be enrolled in the Treatment phase. The Treatment Phase is a randomized, double-blind, double dummy, placebo- and active controlled, 5 treatment, 10-sequence, 5 period crossover, single-dose, Williams square design study in healthy male and/or female adult, non drug-dependent recreational users. On Day 1 of each of the Treatment Phase 5 periods, which will be separated by a washout of at least 14 days, participants will receive an oral dose of either NEURONTIN® 1800 mg, 1200 mg or 600 mg or 20 mg diazepam, or placebo. Study treatments will be administered under fasted conditions (overnight fast and no food until 4 hours after dosing). Water will be allowed without restriction until 1 hour prior to dosing and 1 hour after dosing.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female participants must be 18 to 65 years of age, inclusive, at the time of screening.
2. Participants must meet reproductive criteria as outlined in the protocol.
3. Male and female participants who are overtly healthy. Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, complete physical examination, vital signs, 12-lead electrocardiogram (ECG), and/or clinical laboratory tests.
4. Participants must be recreational sedative users, defined as those reporting using a sedative agent (eg, barbiturates, benzodiazepines) for its intoxicating effects on at least 10 lifetime occasions and at least once in the 12 weeks before the Screening Visit (Visit 1), but who have no signs of dependence and are not seeking treatment for their sedative use.
5. Participants must satisfactorily complete both the Naloxone Challenge and the Drug Discrimination phases.
6. Participants who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, lifestyle considerations, and other study procedures.
7. Body mass index (BMI) of 17.5 to 34 kg/m2, inclusive; and a total body weight >50 kg (110 lb).
8. Capable of giving signed informed consent as described in the protocol, which includes compliance with the requirements and restrictions listed in the informed consent document (ICD) and in this protocol.

Exclusion Criteria

1. Participants with current or past diagnosis of any type of drug dependence within the past year. Diagnosis of substance and/or alcohol dependence (excluding caffeine and nicotine) will be assessed by the Investigator using the Diagnostic and Statistical Manual of Mental Disorders IV (DSM-IV) criteria performed at Screening. Current drug use will be allowed if the candidate can produce a negative urine sample and are free of any signs/symptoms of withdrawal. The candidate will be informed if they have a positive breathalyzer test.
2. Participants are heavy smokers or users of other types of nicotine products (>20 cigarettes equivalents per day)
3. Participants are unable to abstain from smoking for at least 2 hours before and at least 8 hours after study drug administration.
4. Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
5. Participants with any history of sleep apnea, myasthenia or glaucoma.
6. Any condition possibly affecting drug absorption (eg, gastrectomy) excluding cholecystectomy within 1 year prior to study.
7. Clinical or laboratory evidence of active hepatitis A infection or a history of human immunodeficiency virus (HIV) infection, hepatitis B, or hepatitis C, and/or positive testing for HIV, hepatitis B surface antigen (HBsAg), hepatitis B core antibody (HBcAb), or hepatitis C antibody (HCVAb).
8. Participants with active suicidal ideation or suicidal behavior within 5 year prior to Screening as determined through the use of the Columbia-Suicide Severity Rating Scale (C-SSRS) or active ideation identified at Screening or on Day -1.
9. Other acute or chronic medical or psychiatric condition including recent (within the past year) or active suicidal ideation or behavior or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the participant inappropriate for entry into this study.
10. Use of prescription or nonprescription drugs and dietary supplements within 7 days or 5 half-lives (whichever is longer) prior to the first dose of investigational product. (Refer to Section 6.5 for additional details).
11. Herbal supplements and herbal medications must be discontinued at least 28 days prior to the first dose of study medication.
12. Previous administration with an investigational drug within 30 days (or as determined by the local requirement) or 5 half-lives (whichever is longer) preceding the first dose of investigational product used in this study.
13. Positive urine drug screen (UDS) for substances of abuse at each admission in Qualification and Treatment Phase, excluding tetrahydrocannabinol (THC). If a participant presents with a positive UDS excluding THC at any admission or any visit, the investigator, at his/her discretion, may reschedule a repeat UDS until the UDS is negative, excluding THC, before the participant is permitted to participate in any phase of the study.
14. Participants unable to abstain from using THC during the Qualification and Treatment Phases of the study..
15. Has participated in, is currently participating in, or is seeking treatment for substance-and/or alcohol-related disorders (excluding nicotine and caffeine).
16. Has a positive alcohol breathalyzer test at Screening or upon admission to the study center at Visits 2-6. Positive results may be repeated and/or participants re-scheduled at the Investigator's discretions.
17. Screening sitting BP >=140 mm Hg (systolic) or >=90 mm Hg (diastolic), following at least 5 minutes of rest. If BP is >=140 mm Hg (systolic) or >=90 mm Hg (diastolic), the BP should be repeated 2 more times and the average of the 3 BP values should be used to determine the participant's eligibility. Repeated BP tests should be spaced at least 5 minutes apart.
18. Baseline (screening) 12-lead electrocardiogram (ECG) that demonstrates clinically relevant abnormalities that may affect participant safety or interpretation of study results (eg, baseline corrected QT (QTc) interval >450 msec, complete left bundle branch block [LBBB], signs of an acute or indeterminate-age myocardial infarction, ST-T interval changes suggestive of myocardial ischemia, second- or third-degree atrioventricular [AV] block, or serious bradyarrhythmias or tachyarrhythmias). If the baseline uncorrected QT interval is >450 msec, this interval should be rate-corrected using the Fridericia method and the resulting QTcF should be used for decision making and reporting. If QTc exceeds 450 msec, or QRS exceeds 120 msec, the ECG should be repeated 2 more times and the average of the 3 QTc or QRS values should be used to determine the participant's eligibility. Computer-interpreted ECGs should be overread by a physician experienced in reading ECGs before excluding participants.
19. Participants with ANY of the following abnormalities in clinical laboratory tests at screening, as assessed by the study-specific laboratory and confirmed by a single repeat test, if deemed to be clinically significant in the opinion of the investigator:

    * Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) level >=1.5 × upper limit of normal (ULN);
    * Total bilirubin level >=1.5 × ULN; participants with a history of Gilbert's syndrome may have direct bilirubin measured and would be eligible for this study provided the direct bilirubin level is <= ULN.
20. Blood donation (excluding plasma donations) of approximately 1 pint (500 mL) or more within 60 days prior to dosing.
21. History of sensitivity to heparin or heparin-induced thrombocytopenia.
22. Unwilling or unable to comply with the criteria in the Lifestyle Considerations section of this protocol.
23. History of hypersensitivity to gabapentin or diazepam or any of the components in the formulation of the study products.
24. Investigator site staff members directly involved in the conduct of the study and their family members, site staff members otherwise supervised by the investigator, or Sponsor employees, including their family members, directly involved in the conduct of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2021-03-29 (Actual); Primary Completion 2022-11-10 (Actual); Study Completion 2022-11-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Pharmaceutical Research Associates, Inc., Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Subjects entered a Qualification phase involving a naloxone challenge test (to exclude subjects who were opioid dependent) and a drug discrimination test (to confirm they can tell the difference between diazepam and placebo). Only subjects who passed the tests in the Qualification phase were randomized into the Treatment phase where they received the 5 different single dose study treatments, each separated by a washout of at least 14 days, in the order specified for Sequences 1-10 below
Groups:
- Sequence 1: Period 1 Gabapentin 600 mg - Period 2 Gabapentin 1200 mg - Period 3 Placebo - Period 4 Gabapentin 1800 mg - Period 5 Diazepam 20 mg
- Sequence 2: Period 1 Gabapentin 600 mg - Period 2 Placebo - Period 3 Gabapentin 1200 mg - Period 4 Diazepam 20 mg - Period 5 Gabapentin 1800 mg
- Sequence 3: Period 1 Gabapentin 1200 mg - Period 2 Gabapentin 600 mg - Period 3 Gabapentin 1800 mg - Period 4 Placebo - Period 5 Diazepam 20 mg
- Sequence 4: Period 1 Gabapentin 1200 mg - Period 2 Gabapentin 1800 mg - Period 3 Gabapentin 600 mg - Period 4 Diazepam 20 mg - Period 5 Placebo
- Sequence 5: Period 1 Gabapentin 1800 mg - Period 2 Gabapentin 1200 mg - Period 3 Diazepam 20 mg - Period 4 Gabapentin 600 mg - Period 5 Placebo
- Sequence 6: Period 1 Gabapentin 1800 mg - Period 2 Diazepam 20 mg - Period 3 Gabapentin 1200 mg - Period 4 Placebo - Period 5 Gabapentin 600 mg
- Sequence 7: Period 1 Diazepam 20 mg - Period 2 Gabapentin 1800 mg - Period 3 Placebo - Period 4 Gabapentin 1200 mg - Period 5 Gabapentin 600 mg
- Sequence 8: Period 1 Diazepam 20 mg - Period 2 Placebo - Period 3 Gabapentin 1800 mg - Period 4 Gabapentin 600 mg - Period 5 Gabapentin 1200 mg
- Sequence 9: Period 1 Placebo - Period 2 Gabapentin 600 mg - Period 3 Diazepam 20 mg - Period 4 Gabapentin 1200 mg -Period 5 Gabapentin 1800 mg
- Sequence 10: Period 1 Placebo - Period 2 Diazepam 20 mg - Period 3 Gabapentin 600 mg - Period 4 Gabapentin 1800 mg - Period 5 Gabapentin 1200 mg
Period: Overall Study
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6 | Sequence 7 | Sequence 8 | Sequence 9 | Sequence 10
Started | 5 | 5 | 6 | 5 | 5 | 5 | 6 | 5 | 5 | 5
Completed | 4 | 5 | 5 | 5 | 5 | 5 | 6 | 5 | 5 | 5
Not Completed | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who completed all 5 treatment periods of the Treatment Phase, excluding those subjects who had scores for the primary endpoint (maximum Drug Liking Visual Analog Scale score) that were within 5 points across all 5 treatments and/or had high placebo scores for the primary endpoint (maximum Drug Liking Visual Analog Scale score for placebo was > 60 on a 100 point scale and the primary endpoint for placebo was 5 or more points greater than that for the positive control, diazepam)
Groups:
- Modified Completer Population: All participants who completed all 5 treatment periods of the Treatment Phase but excluding those subjects who had scores for the primary endpoint (maximum Drug Liking Visual Analog Scale score) that were within 5 points across all 5 treatments and/or had high placebo scores for the primary endpoint (maximum Drug Liking Visual Analog Scale score for placebo was > 60 on a 100 point scale and the primary endpoint for placebo was 5 or more points greater than that for the positive control, diazepam). This was the primary analysis population.
Arm/Group | Modified Completer Population
Number analyzed (Participants) | 41
Age, Continuous [Mean (Standard Deviation); unit: Years] | 34.2 (9.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 35
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 12
  White | 25
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 41

OUTCOME MEASURES:

1. Primary Outcome: Bipolar Visual Analog Scale (VAS) for "Drug Liking" Maximum Effect (Emax).
Description: Drug liking assesses how much a participant likes or dislikes a drug effect at the time the question is being asked. It is scored using a 100 mm visual analogue scale (VAS), where 0 mm = "Strong Disliking", 50 mm = "Neither Like nor Dislike", and 100 mm = "Strong Liking"
Time Frame: up to 72 hours after treatments
Population: Modified completer population
Measure: Mean (Standard Error); unit: Score on a scale
Groups:
- Placebo: single dose
  placebo: participants received a single oral dose of placebo
- Diazepam 20 mg: single dose
  diazepam 20 mg: participants received a single oral dose of 20 mg dose of diazepam
- Gabapentin 600 mg: single dose
  gabapentin 600 mg: participants received a single oral dose of gabapentin 600 mg
- Gabapentin 1200 mg: single dose
  gabapentin 1200 mg: participants received a single oral dose of gabapentin 1200 mg
- Gabapentin 1800 mg: single dose
  gabapentin 1800 mg: participants received a single oral dose of gabapentin 1800 mg
Arm/Group | Placebo | Diazepam 20 mg | Gabapentin 600 mg | Gabapentin 1200 mg | Gabapentin 1800 mg
Number analyzed (Participants) | 41 | 41 | 41 | 41 | 41
Score on a scale | 51.98 (0.955) | 79.37 (2.533) | 61.95 (2.418) | 61.39 (2.209) | 60.95 (2.270)
Statistical Analysis 1: Comparison: Placebo vs Diazepam 20 mg; The sensitivity and integrity of the study was validated by comparing the mean responses of diazepam, the positive control (C), to the placebo (P): H0: μC - μP ≤ δ1 versus Ha: μC - μP > δ1 where δ1 = 15; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = 30.9, 95% CI 1-sided [lower limit 26.2], Standard Error of Mean 2.85
Statistical Analysis 2: Comparison: Placebo vs Gabapentin 600 mg; The primary analysis evaluated whether gabapentin (T) produced mean responses that show abuse potential similar to placebo. H0: μT - μP ≥ δ3 versus Ha: μT - μP < δ3 where δ3 =11; Test type: Non-Inferiority — Non-inferiority margin = 11; p = 0.3581, Mixed Models Analysis; Mean Difference (Final Values) = 10.0, 95% CI 1-sided [upper limit 14.7], Standard Error of Mean 2.84
Statistical Analysis 3: Comparison: Placebo vs Gabapentin 1200 mg; [analysis description as in outcome 1, analysis 2]; Test type: Non-Inferiority — Non-inferiority margin = 11; p = 0.3051, Mixed Models Analysis; Mean Difference (Final Values) = 9.5, 95% CI 1-sided [upper limit 14.3], Standard Error of Mean 2.85
Statistical Analysis 4: Comparison: Placebo vs Gabapentin 1800 mg; [analysis description as in outcome 1, analysis 2]; Test type: Non-Inferiority — Non-inferiority margin = 11; p = 0.2179, Mixed Models Analysis; Mean Difference (Final Values) = 8.8, 95% CI 1-sided [upper limit 13.5], Standard Error of Mean 2.83
Statistical Analysis 5: Comparison: Diazepam 20 mg vs Gabapentin 600 mg; The null and alternative hypotheses for evaluating whether gabapentin (T) produced mean responses that show less abuse potential than diazepam (C) were: H0: μC - μT ≤ δ2 versus Ha: μC - μT > δ2 where δ2 =0; Test type: Non-Inferiority — Non-inferiority margin = 0; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = 20.9, 95% CI 1-sided [lower limit 16.3], Standard Error of Mean 2.84
Statistical Analysis 6: Comparison: Diazepam 20 mg vs Gabapentin 1200 mg; [analysis description as in outcome 1, analysis 5]; Test type: Non-Inferiority — Non-inferiority margin = 0; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = 21.4, 95% CI 1-sided [lower limit 16.7], Standard Error of Mean 2.84
Statistical Analysis 7: Comparison: Diazepam 20 mg vs Gabapentin 1800 mg; [analysis description as in outcome 1, analysis 5]; Test type: Non-Inferiority — Non-inferiority margin = 0; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = 22.1, 95% CI 1-sided [lower limit 17.4], Standard Error of Mean 2.85

2. Secondary Outcome: Bipolar VAS for "Drug Liking" (Time for Maximum Effect, Emax [TEmax])
Description: Time after dosing when the maximum effect for Drug Liking VAS is reached
Time Frame: up to 72 hours after treatments
Population: Modified completer population
Measure: Median (Full Range); unit: Hours
Groups:
- Placebo: Participants received a single oral dose of placebo
- Diazepam 20 mg: Participants received a single oral dose of 20 mg dose of diazepam
- Gabapentin 600 mg: Participants received a single oral dose of gabapentin 600 mg
- Gabapentin 1200 mg: Participants received a single oral dose of gabapentin 1200 mg
- Gabapentin 1800 mg: Participants received a single oral dose of gabapentin 1800 mg
Arm/Group | Placebo | Diazepam 20 mg | Gabapentin 600 mg | Gabapentin 1200 mg | Gabapentin 1800 mg
Number analyzed (Participants) | 41 | 41 | 41 | 41 | 41
Hours | 0.2 [0.2 to 72] | 1.51 [0.2 to 8.0] | 2.0 [0.2 to 48.0] | 2.0 [0.2 to 12.0] | 2.5 [0.2 to 12.0]

3. Secondary Outcome: Bipolar VAS for "Drug Liking" (Area Under the Effect-time Profile From Time 0 to the Time of the Last Quantifiable Concentration [AUEClast])
Description: Area under the effect-time profile from time 0 to the time of the last available data for the "Drug liking" visual analog scale which assesses how much a participant likes or dislikes a drug effect at the time the question ("at this moment, my liking this drug is") is being asked. It is scored using a 100 mm visual analogue scale (VAS), where 0 mm = "Strong Disliking", 50 mm = "Neither Like nor Dislike", and 100 mm = "Strong Liking". The minimum and maximum possible scores are approximately 0 and 7200 if a subject scores 0 mm (strong disliking) and 100 mm (strong liking) respectively at every timepoint up to 72 hours.
Time Frame: Up to 72 hours after treatments (Assessments were made at the following timepoints after each treatment: 0, 0.25, 0.5,1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 24, 36, 48, and 72 hours)
Population: Modified completer population
Measure: Mean (Standard Error); unit: units on a scale * hour
Arm/Group | Placebo | Diazepam 20 mg | Gabapentin 600 mg | Gabapentin 1200 mg | Gabapentin 1800 mg
Number analyzed (Participants) | 41 | 41 | 41 | 41 | 41
units on a scale * hour | 3441.77 (101.695) | 3778.02 (124.372) | 3588.67 (107.642) | 3601.72 (46.538) | 3652.27 (114.555)
Statistical Analysis 1: Comparison: Placebo vs Diazepam 20 mg; Test type: Other; p = 0.0023, Mixed Models Analysis; Mean Difference (Final Values) = 325.8, 90% CI 1-sided [lower limit 138.2], Standard Error of Mean 113.38
Statistical Analysis 2: Comparison: Placebo vs Gabapentin 600 mg; Test type: Other; p = 0.2157, Mixed Models Analysis; Mean Difference (Final Values) = 140.5, 90% CI 2-sided [-82.7 to 363.7], Standard Error of Mean 113.01
Statistical Analysis 3: Comparison: Placebo vs Gabapentin 1200 mg; Test type: Other; p = 0.1720, Mixed Models Analysis; Mean Difference (Final Values) = 155.4, 90% CI 2-sided [-68.3 to 379.1], Standard Error of Mean 113.25
Statistical Analysis 4: Comparison: Placebo vs Gabapentin 1800 mg; Test type: Other; p = 0.0622, Mixed Models Analysis; Mean Difference (Final Values) = 212.2, 90% CI 2-sided [-11.0 to 435.5], Standard Error of Mean 113.01
Statistical Analysis 5: Comparison: Diazepam 20 mg vs Gabapentin 600 mg; Test type: Other; p = 0.1031, Mixed Models Analysis; Mean Difference (Final Values) = -185, 90% CI 2-sided [-409 to 37.94], Standard Error of Mean 113.04
Statistical Analysis 6: Comparison: Diazepam 20 mg vs Gabapentin 1200 mg; Test type: Other; p = 0.1334, Mixed Models Analysis; Mean Difference (Final Values) = -170, 90% CI 2-sided [-394 to 52.71], Standard Error of Mean 112.97
Statistical Analysis 7: Comparison: Diazepam 20 mg vs Gabapentin 1800 mg; Test type: Other; p = 0.3189, Mixed Models Analysis; Mean Difference (Final Values) = -114, 90% CI 2-sided [-338 to 110.8], Standard Error of Mean 113.59

4. Secondary Outcome: Unipolar VAS for "High" (Maximum Effect, Emax)
Description: Maximum effect on the 100 mm visual analog scale for the question "I am feeling high" where 0 = "not at all" and 100 ="extremely"
Time Frame: up to 72 hours after treatments
Population: Modified completer population
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | Diazepam 20 mg | Gabapentin 600 mg | Gabapentin 1200 mg | Gabapentin 1800 mg
Number analyzed (Participants) | 41 | 41 | 41 | 41 | 41
Score on a scale | 5.80 (2.272) | 61.56 (5.056) | 23.02 (4.351) | 26.93 (4.717) | 27.66 (4.753)
Statistical Analysis 1: Comparison: Placebo vs Diazepam 20 mg; Test type: Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = 55.77, 90% CI 1-sided [lower limit 46.89], Standard Error of Mean 5.362
Statistical Analysis 2: Comparison: Placebo vs Gabapentin 600 mg; Test type: Other; p = 0.0016, Mixed Models Analysis; Mean Difference (Final Values) = 17.18, 90% CI 2-sided [6.61 to 27.74], Standard Error of Mean 5.348
Statistical Analysis 3: Comparison: Placebo vs Gabapentin 1200 mg; Test type: Other; p = 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = 21.38, 90% CI 2-sided [10.79 to 31.96], Standard Error of Mean 5.360
Statistical Analysis 4: Comparison: Placebo vs Gabapentin 1800 mg; Test type: Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = 22.50, 90% CI 2-sided [11.92 to 33.07], Standard Error of Mean 5.352
Statistical Analysis 5: Comparison: Diazepam 20 mg vs Gabapentin 600 mg; Test type: Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -38.6, 90% CI 2-sided [-49.1 to -28.1], Standard Error of Mean 5.312
Statistical Analysis 6: Comparison: Diazepam 20 mg vs Gabapentin 1200 mg; Test type: Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -34.4, 90% CI 2-sided [-44.9 to -23.9], Standard Error of Mean 5.308
Statistical Analysis 7: Comparison: Diazepam 20 mg vs Gabapentin 1800 mg; Test type: Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -33.3, 90% CI 2-sided [-43.8 to -22.7], Standard Error of Mean 5.337

5. Secondary Outcome: Unipolar VAS for "High" (Time for Maximum Effect, Emax [TEmax])
Description: Time after dosing when the maximum effect for "High" VAS is reached
Time Frame: up to 72 hours after treatments
Population: Modified completer population
Measure: Median (Full Range); unit: Hours
Arm/Group | Placebo | Diazepam 20 mg | Gabapentin 600 mg | Gabapentin 1200 mg | Gabapentin 1800 mg
Number analyzed (Participants) | 41 | 41 | 41 | 41 | 41
Hours | 0.20 [0.2 to 6.0] | 1.96 [0.2 to 6.0] | 1.50 [0.2 to 8.0] | 2.00 [0.2 to 8.0] | 2.50 [0.2 to 24.0]

6. Secondary Outcome: Unipolar VAS for "High" (Area Under the Effect-time Profile From Time 0 to the Time of the Last Quantifiable Concentration [AUEClast])
Description: Area under the effect-time profile from time 0 to the time of the last available data for the "High" visual analog scale which measures on a 100 mm visual analog scale the subject's response to the question "I am feeling high" where 0 ="not at all" and 100 ="extremely". The minimum and maximum possible scores are 0 and approximately 7200 if a subject scores 0 mm (not at all) and 100 mm (extremely) respectively at every timepoint up to 72 hours.
Time Frame: as for outcome 3
Population: Modified completer population
Measure: Mean (Standard Error); unit: units on a scale * hour
Arm/Group | Placebo | Diazepam 20 mg | Gabapentin 600 mg | Gabapentin 1200 mg | Gabapentin 1800 mg
Number analyzed (Participants) | 41 | 41 | 41 | 41 | 41
units on a scale * hour | 15.06 (5.993) | 250.38 (40.596) | 83.08 (23.583) | 112.74 (39.041) | 109.07 (24.600)
Statistical Analysis 1: Comparison: Placebo vs Diazepam 20 mg; Test type: Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = 234.9, 90% CI 1-sided [lower limit 171.7], Standard Error of Mean 38.174
Statistical Analysis 2: Comparison: Placebo vs Gabapentin 600 mg; Test type: Other; p = 0.0834, Mixed Models Analysis; Mean Difference (Final Values) = 66.30, 90% CI 2-sided [-8.86 to 141.5], Standard Error of Mean 38.048
Statistical Analysis 3: Comparison: Placebo vs Gabapentin 1200 mg; Test type: Other; p = 0.0103, Mixed Models Analysis; Mean Difference (Final Values) = 99.06, 90% CI 2-sided [23.75 to 174.4], Standard Error of Mean 38.128
Statistical Analysis 4: Comparison: Placebo vs Gabapentin 1800 mg; Test type: Other; p = 0.0116, Mixed Models Analysis; Mean Difference (Final Values) = 97.20, 90% CI 2-sided [22.05 to 172.4], Standard Error of Mean 38.048
Statistical Analysis 5: Comparison: Diazepam 20 mg vs Gabapentin 600 mg; Test type: Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -169, 90% CI 2-sided [-244 to -93.4], Standard Error of Mean 38.060
Statistical Analysis 6: Comparison: Diazepam 20 mg vs Gabapentin 1200 mg; Test type: Other; p = 0.0005, Mixed Models Analysis; Mean Difference (Final Values) = -136, 90% CI 2-sided [-211 to -60.7], Standard Error of Mean 38.036
Statistical Analysis 7: Comparison: Diazepam 20 mg vs Gabapentin 1800 mg; Test type: Other; p = 0.0004, Mixed Models Analysis; Mean Difference (Final Values) = -138, 90% CI 2-sided [-213 to -62.2], Standard Error of Mean 38.243

7. Secondary Outcome: Bipolar VAS for "Take Drug Again" at 24 Hour Post Dose
Description: 100 mm visual analog scale for the question "I would take this drug again" where 0 ="definitely not", 50 = "neutral", and 100 = "definitely so".
Time Frame: At 24 hours after treatment
Population: Modified completer population
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | Diazepam 20 mg | Gabapentin 600 mg | Gabapentin 1200 mg | Gabapentin 1800 mg
Number analyzed (Participants) | 41 | 41 | 41 | 41 | 41
Score on a scale | 48.66 (1.955) | 63.10 (3.218) | 58.28 (2.453) | 55.63 (2.318) | 54.90 (2.773)

8. Secondary Outcome: Bipolar VAS for "Take Drug Again" at 36 Hour Post Dose
Description: as for outcome 7
Time Frame: At 36 hours after treatment
Population: Modified completer population
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | Diazepam 20 mg | Gabapentin 600 mg | Gabapentin 1200 mg | Gabapentin 1800 mg
Number analyzed (Participants) | 41 | 41 | 41 | 41 | 41
Score on a scale | 49.27 (1.392) | 64.95 (2.846) | 55.33 (2.546) | 55.73 (1.988) | 54.93 (2.403)

9. Secondary Outcome: Bipolar VAS for "Take Drug Again" at 48 Hour Post Dose
Description: as for outcome 7
Time Frame: At 48 hours after treatment
Population: Modified completer population
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | Diazepam 20 mg | Gabapentin 600 mg | Gabapentin 1200 mg | Gabapentin 1800 mg
Number analyzed (Participants) | 41 | 41 | 41 | 41 | 41
Score on a scale | 49.24 (1.390) | 62.24 (3.232) | 55.90 (1.954) | 52.80 (1.785) | 53.59 (2.150)

10. Secondary Outcome: Bipolar VAS for "Take Drug Again" at 72 Hour Post Dose
Description: as for outcome 7
Time Frame: At 72 hours after treatment
Population: Modified completer population
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | Diazepam 20 mg | Gabapentin 600 mg | Gabapentin 1200 mg | Gabapentin 1800 mg
Number analyzed (Participants) | 41 | 41 | 41 | 41 | 41
Score on a scale | 49.17 (1.402) | 63.88 (3.679) | 55.90 (1.921) | 53.76 (2.583) | 54.46 (2.184)

11. Secondary Outcome: Bipolar VAS for "Overall Drug Liking" at 24 Hour Post Dose
Description: 100 mm visual analog scale for the question "Overall, my liking for this drug is" where0 = "definitely not", 50 = "neutral", and 100 = "definitely so".
Time Frame: At 24 hours after treatment
Population: Modified completer population
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | Diazepam 20 mg | Gabapentin 600 mg | Gabapentin 1200 mg | Gabapentin 1800 mg
Number analyzed (Participants) | 41 | 41 | 41 | 41 | 41
Score on a scale | 48.20 (1.909) | 63.66 (3.578) | 57.10 (2.560) | 54.15 (2.618) | 53.90 (2.602)

12. Secondary Outcome: Bipolar VAS for "Overall Drug Liking" at 36 Hour Post Dose
Description: as for outcome 11
Time Frame: At 36 hours after treatment
Population: Modified completer population
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | Diazepam 20 mg | Gabapentin 600 mg | Gabapentin 1200 mg | Gabapentin 1800 mg
Number analyzed (Participants) | 41 | 41 | 41 | 41 | 41
Score on a scale | 49.59 (1.584) | 61.83 (2.962) | 54.75 (2.952) | 55.63 (1.757) | 53.49 (2.109)

13. Secondary Outcome: Bipolar VAS for "Overall Drug Liking" at 48 Hour Post Dose
Description: as for outcome 11
Time Frame: At 48 hours after treatment
Population: Modified completer population
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | Diazepam 20 mg | Gabapentin 600 mg | Gabapentin 1200 mg | Gabapentin 1800 mg
Number analyzed (Participants) | 41 | 41 | 41 | 41 | 41
Score on a scale | 49.68 (1.467) | 61.07 (2.992) | 54.83 (2.485) | 54.66 (2.156) | 53.37 (2.107)

14. Secondary Outcome: Bipolar VAS for "Overall Drug Liking" at 72 Hour Post Dose
Description: as for outcome 11
Time Frame: At 72 hours after treatment
Population: Modified completer population
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | Diazepam 20 mg | Gabapentin 600 mg | Gabapentin 1200 mg | Gabapentin 1800 mg
Number analyzed (Participants) | 41 | 41 | 41 | 41 | 41
Score on a scale | 49.56 (1.503) | 61.46 (3.449) | 55.68 (2.117) | 55.10 (2.222) | 53.46 (2.606)

15. Secondary Outcome: Cmax of Gabapentin
Description: Maximum plasma concentration (Cmax) of gabapentin
Time Frame: Up to 72 hours after treatments (concentrations were measured at the following timepoints after each treatment for this outcome measure: 0, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 24, 36, 48, and 72 hours)
Population: Pharmacokinetic population: all enrolled participants who received study medication and have pharmacokinetic data for the parameters of interest.
Measure: Mean (Standard Deviation); unit: nanograms/milliliter
Arm/Group | Gabapentin 600 mg | Gabapentin 1200 mg | Gabapentin 1800 mg
Number analyzed (Participants) | 52 | 52 | 51
nanograms/milliliter | 4223.47 (1048.963) | 6106.90 (1355.048) | 7373.15 (1874.185)

16. Secondary Outcome: Tmax of Gabapentin
Description: Time when the maximum concentration of gabapentin is reached
Time Frame: Up to 72 hours after treatments (concentrations were measured at the following timepoints after each treatment for thisoutcome measure: 0, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 24, 36, 48 and 72 hours)
Population: as for outcome 15
Measure: Median (Full Range); unit: Hours
Arm/Group | Gabapentin 600 mg | Gabapentin 1200 mg | Gabapentin 1800 mg
Number analyzed (Participants) | 52 | 52 | 51
Hours | 2.78 [1.0 to 6.1] | 2.55 [1.0 to 6.1] | 2.55 [1.0 to 6.1]

17. Secondary Outcome: AUClast of Gabapentin
Description: Area under the effect time profile from time 0 to the time of the last quantifiable concentration (AUClast) of gabapentin
Time Frame: up to 72 hours after treatment (concentrations were measured at the following timepoints after each treatment for thisoutcome measure: 0, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 24, 36, 48 and 72 hours)
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: nanograms*hour/milliliter
Arm/Group | Gabapentin 600 mg | Gabapentin 1200 mg | Gabapentin 1800 mg
Number analyzed (Participants) | 52 | 52 | 51
nanograms*hour/milliliter | 41848.88 (10659.677) | 66972.60 (15921.032) | 80483.05 (22369.826)

18. Secondary Outcome: Terminal Half-life of Gabapentin
Description: Terminal half-life (t½) of gabapentin
Time Frame: as for outcome 17
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Gabapentin 600 mg | Gabapentin 1200 mg | Gabapentin 1800 mg
Number analyzed (Participants) | 51 | 52 | 50
Hours | 7.69 (2.496) | 13.83 (12.988) | 14.43 (11.130)

ADVERSE EVENTS:
Time Frame: During the entire Treatment Phase of the study, which encompassed the time interval from admission of the subject to their first Treatment Period until 28 days after study drug dosing in their last (6th) Treatment Period, including the washout in between. The total duration of the Treatment Phase for each subject was dependent on visit scheduling and whether the subject completed treatment periods, and it lasted up to approximately 13 weeks.
Description: Adverse events that occur during the washout interval between treatment visits or during the follow up after the final study drug dosing counted under the previous treatment visit
Arm/Group | Placebo | Diazepam 20 mg | Gabapentin 600 mg | Gabapentin 1200 mg | Gabapentin 1800 mg
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/50 | 0/52 | 0/52 | 0/51
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50 | 0/52 | 0/52 | 0/51
Other Adverse Events (participants affected / at risk) | 11/50 | 30/50 | 20/52 | 24/52 | 23/51
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=50) | Diazepam 20 mg (N=50) | Gabapentin 600 mg (N=52) | Gabapentin 1200 mg (N=52) | Gabapentin 1800 mg (N=51)
Somnolence (Nervous system disorders) | 2 (2) | 15 (15) | 7 (7) | 8 (8) | 10 (10)
Lethargy (Nervous system disorders) | 2 (2) | 6 (6) | 4 (4) | 2 (2) | 2 (2)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1) | 5 (5) | 5 (5)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 4 (4) | 3 (3)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Fatigue (General disorders) | 1 (1) | 5 (5) | 3 (3) | 4 (4) | 2 (2)
Feeling of relaxation (General disorders) | 2 (2) | 4 (4) | 3 (3) | 0 (0) | 2 (2)
Euphoric mood (Psychiatric disorders) | 1 (1) | 6 (6) | 6 (6) | 5 (5) | 4 (4)
Sedation (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Cognitive idsorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Scleral disorder (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Visual impairment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diplopia (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SARS-CoV-2 test positive (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-04-29): https://cdn.clinicaltrials.gov/large-docs/36/NCT04570436/Prot_000.pdf
  • Statistical Analysis Plan (2023-01-27): https://cdn.clinicaltrials.gov/large-docs/36/NCT04570436/SAP_001.pdf